CLINICAL TRIAL: NCT06941922
Title: Testicular Evaluation of Azoospermia Using Micro-Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Paul Shin (Other)
Collaborators: Exact Imaging (Industry)
Responsible Party: Sponsor-Investigator, Paul Shin, Principal Study Investigator, Shady Grove Fertility Reproductive Science Center
Organization: Shady Grove Fertility Reproductive Science Center (Other)
Other Study IDs: SHIN-2024-001
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-04

CONDITIONS: Azoospermia
Keywords: azoospermia, infertility, microultrasound, microdissection
MeSH Terms: conditions — Azoospermia; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Men with azoospermia confirmed based on semen analysis
- Post-vasectomy patients with verified azoospermia after the procedure
- Men pre-vasectomy with proven natural fertility or with normal semen analysis

SUMMARY:
The investigation is a small feasibility study to determine whether there are imaging features related to the seminiferous tubules in the testes under microultrasound. The results from this study will provide guidance on the design and power analysis of future studies in this area.

DETAILED DESCRIPTION:
Currently available ultrasound (US) technology is approximately 12 MHz and offers enough resolution to determine the presence of a tumor or varicocele, but has no real predictive value in terms of imaging robust seminiferous tubules. MicroUS offers significantly higher resolution - down to 70 microns. The average width of a normal seminiferous tubule is 200-250 microns. (Amer 1837). The average width of an atrophic SCO tubule is 75 microns. This echotexture difference cannot be visualized by a conventional ultrasound scan but should, in theory, be detected by a higher resolution (higher MHz) microUS scan.

This is a feasibility study to image 40 azoospermic or healthy controls in order to determine whether microultrasound (microUS) images can visualize differences within the testes of these subjects which may be useful in diagnosing the cause of azoospermia and regional differences within the testes where sperm retrieval may be more effective.

Specifically, in men with obstructive azoospermia we expect to visualize normal seminiferous tubules while in men with non-obstructive azoospermia we expect to visualize both normal and atrophic seminiferous tubules.

The normal tubules in cases of obstructive azoospermia will act as a control by providing an example of normal imaging within a closely related population. Localization of normal tubules within the NOA (non-obstructive azoospermia) population may simplify the microTESE procedure by reducing the amount of dissection required. Additionally, the ability to predict the success of the procedure (i.e. presence of normal tubules) would improve risk/benefit decision-making for men considering it.

ELIGIBILITY:
Inclusion criteria:

1. Men with azoospermia confirmed based on semen analysis
2. Post-vasectomy patients with verified azoospermia after the procedure
3. Men pre-vasectomy with proven natural fertility or with normal semen analysis
4. Males assigned at birth over the age of 18

Exclusion criteria:

1. History of prior microdissection of the testes
2. History of hypogonadotropic hypogonadism

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who make sperm
Study Population: Participants who meet inclusion and exclusion criteria and have been referred to the study infertility clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The micro-ultrasound imaging procedure produces imaging features which correlate to the presence of sperm within the seminiferous tubules of the testes | From time of enrollment to end of scanning (45 minutes)
  The investigation is a small feasibility study to determine whether there are imaging features related to the seminiferous tubules in the testes under microUS. The results from this study will provide guidance on the design and power analysis of future studies in this area.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Shin, MD, Principal Investigator — Shady Grove Fertility
Locations (2):
- Shady Grove Fertility, Rockville, Maryland, United States
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided